CLINICAL TRIAL: NCT04250402
Title: The Incidence Risks of Gallstones After Radical Surgery in Different Types of Gastric Cancer
Brief Title: The Incidence of Gallstones After Gastric Cancer Surgery
Status: Completed | Type: Observational
Sponsor: Hepatopancreatobiliary Surgery Institute of Gansu Province (Other)
Responsible Party: Principal Investigator, Wenbo Meng, Direct of surgery, Hepatopancreatobiliary Surgery Institute of Gansu Province
Other Study IDs: Gallstones after gastrectomy
Record Dates: First submitted 2020-01-29; First posted 2020-01-31 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Gallstones; Gastric Cancer
Keywords: Gallstones; Gastric cancer; Gastrectomy; ESD; Vagus nerve
MeSH Terms: conditions — Gallstones; Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Arm 1: Endoscopic submucosal dissection. Endoscopic submucosal dissection is an endoscopic procedure which can achieve en bloc resection of GI tumor. ESD is characterized by three steps: injecting fluid into the submucosa to elevate the lesion from the muscle layer, circumferential cutting of the surrounding mucosa of the lesion, and subsequent dissection of the connective tissue of the submucosa beneath the lesion. The ESD procedure will be carried out by experienced endoscopists.
  Other Name: ESD
  Interventions: Procedure: Resection
- Arm 2: Distal subtotal gastrectomy with D2 lymphadenectomy. After exclusion of T4b, bulky lymph nodes, or distant metastasis case, distal subtotal gastrectomy and D2 lymph node dissection will be performed with curative treated intent.
  The type of reconstruction will be selected according to the surgeon's experience and anastomotic procedure is performed extracorporeally.
  Interventions: Procedure: Resection
- Arm 3: Total gastrectomy with D2 lymphadenectomy will be performed with curative treated intent. The type of reconstruction will be with jejunal interposition reconstruction.
  Interventions: Procedure: Resection
- Arm 4: Proximal gastrectomy with D2 lymphadenectomy. The type of reconstruction will be jejunal interposition with double anastomosis method.
  Interventions: Procedure: Resection

INTERVENTIONS:
Procedure: Resection — Radical resection.

SUMMARY:
Through previous clinical observations and literature, we found that the incidence of gallstones in patients after gastric cancer radical resection was significantly higher than that in the normal population (4%). However, its pathogenesis has not been clarified. We compare the risk of gallbladder stones after four different radical gastric cancer surgical methods, in order to provide prevention and treatment strategies for people with gallstones after gastric cancer.

DETAILED DESCRIPTION:
A large number of clinical studies have found that the incidence of gallstones in patients with radical gastric cancer is higher than that in the normal population. However, its pathogenesis has not been clarified, and there is still controversy about the prophylactic removal of gallbladder in patients with gastric cancer. The investigator's previous study found that there was no statistical difference in the incidence of gallstones after laparoscopic distal gastrectomy (LDG), laparoscopic total gastrectomy (LTG) and laparoscopic proximal gastrectomy (LPG). A common feature of the three surgical methods is that the vagus nerve were more or less cut during the operation. Therefore, we plan to further collect gastric cancer patients undergoing endoscopic submucosal dissection (ESD) surgery in order to answer whether the vagus nerve cut during surgery will increase the incidence of gallstones.

ELIGIBILITY:
Inclusion Criteria:

* Gastric cancer patients
* Age from over 18 to under 75 years

Exclusion Criteria:

* Gallbladder disease before surgery
* Gallbladder has been remove
* History of previous upper abdominal surgery
* History of previous gastrectomy, endoscopic mucosal resection or endoscopic submucosal dissection
* History of other malignant disease within past five years
* History of previous neoadjuvant chemotherapy or radiotherapy
* History of unstable angina or myocardial infarction within past six months
* History of cerebrovascular accident within past six months
* Requirement of simultaneous surgery for other disease
* Emergency surgery due to complication (bleeding, obstruction or perforation) caused by gastric cancer
* Pregnant women or breastfeeding
* Unwillingness or inability to consent for the study
* Severe mental disorder
* Unstable vital signs Coagulation dysfunction (INR>1.5)
* Low peripheral blood platelet count (<50×10 ^9 / L) or using anti- coagulation drugs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Gastric cancer patients
Sampling Method: Probability Sample
Enrollment: 1019 (Actual)
Dates: Start 2020-02-14 (Actual); Primary Completion 2024-11-16 (Actual); Study Completion 2024-11-16 (Actual)

PRIMARY OUTCOMES:
Number of gallstone patients | 3 years
  Four different gastric cancer patients were followed up for more than 1 year. The number of patients with gallbladder stones revealed by B-ultrasound

SECONDARY OUTCOMES:
Number of malignant metastasis | 3 years
  Number of malignant metastases after radical gastrectomy in surgery methods of gastric cancer patients
Number of short-term deaths | 3 months
  Number of short-term deaths after radical gastrectomy in surgery methods of gastric cancer patients
Number of physical regurgitation, nausea, vomiting, diarrhea, constipation | 3 years
  The number of physical regurgitation, nausea, vomiting, diarrhea, constipation, and other events that affect quality of life in four surgery methods of gastric cancer patients

CONTACTS AND LOCATIONS:
Overall Officials: Wenbo Meng, M.D., Ph. D., Principal Investigator — Hepatopancreatobiliary Surgery Institute of Gansu Province
Locations (2):
- China (2):
  - Hepatopancreatobiliary Surgery Institute of Gansu Province, Lanzhou, Gansu
  - Wuwei turmour hospital, Wuwei, Gansu

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Park DJ, Kim KH, Park YS, Ahn SH, Park do J, Kim HH. Risk Factors for Gallstone Formation after Surgery for Gastric Cancer. J Gastric Cancer. 2016 Jun;16(2):98-104. doi: 10.5230/jgc.2016.16.2.98. Epub 2016 Jun 24. PMID 27433395
- [Background] Furukawa H, Ohashi M, Honda M, Kumagai K, Nunobe S, Sano T, Hiki N. Preservation of the celiac branch of the vagal nerve for pylorus-preserving gastrectomy: is it meaningful? Gastric Cancer. 2018 May;21(3):516-523. doi: 10.1007/s10120-017-0776-8. Epub 2017 Nov 10. PMID 29127549